CLINICAL TRIAL: NCT02599571
Title: Effects of Nicotine Reduction on Smoking Behavior in ADHD Smokers
Acronym: ADHDenic
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: sponsor discontinued funding
Sponsor: Duke University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency); University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro00066144; 1R01HD083404 (NIH)
Record Dates: First submitted 2015-11-02; First posted 2015-11-06 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Nicotine Dependence; ADHD
MeSH Terms: conditions — Tobacco Use Disorder; Attention Deficit Disorder with Hyperactivity | interventions — Tobacco Products

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Very low nicotine content cigarettes (Other): Reduced nicotine content cigarettes.
  Interventions: Other: Very low nicotine content cigarettes; Other: Conventional nicotine content cigarettes
- Conventional nicotine content cigarettes (Other): Conventional nicotine content cigarettes.
  Interventions: Other: Very low nicotine content cigarettes; Other: Conventional nicotine content cigarettes

INTERVENTIONS:
Other: Very low nicotine content cigarettes — Cigarettes containing a reduced amount of nicotine
  Other Names: Tobacco; Cigarettes
Other: Conventional nicotine content cigarettes — Cigarettes containing a normal amount of nicotine
  Other Names: Tobacco; Cigarettes

SUMMARY:
The purpose of this study is to investigate the impact of different nicotine levels in cigarettes with individuals who have ADHD.

DETAILED DESCRIPTION:
The purpose of this study is to examine the effects of very low nicotine content (VLNC) cigarettes on smoking behavior, psychiatric symptoms and functioning, and acceptability and adverse outcomes in young adult smokers with ADHD. Participants will attend a screening session, 2 baseline sessions, 6 experimental sessions, and a 30 day follow-up visit. Participants will be asked to smoke only the study cigarettes that we provide for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 40
* Smoke an average of 5-40 cigarettes per day for at least 1 year
* Breath CO levels > 8 ppm (if ≤ 8 ppm, then NicAlert Strip > 6)
* Primary diagnosis of ADHD, any subtype as assessed by the CAADID; T-Score > 65 on one of the DSM- V relevant scales (Inattentive Symptoms, Hyperactive-Impulsive Symptoms, Total Symptoms or ADHD Index) on the Self-Report version of the CAARS; Clinician Rated ADHD-RS score >24.
* Cognitive functioning > 80 as assessed by the KBIT-II

Exclusion Criteria:

* Intention to quit smoking in the next 30 days
* Currently seeking treatment for smoking cessation
* Currently using nicotine replacement therapies or other pharmacotherapies as cessation aid (intermittent use acceptable)
* A quit attempt in the past 30 days resulting in greater than 3 days of abstinence
* Using other tobacco products more than 9 days in the past 30 days
* Significant unstable medical conditions (any significant change in a serious medical condition occurring during the past 3 months including cardiovascular disease, COPD, and cancer, as determined by the study physician at each site)
* Significant unstable psychiatric conditions (any significant change in psychiatric symptoms during the past 3 months as determined by the study physician at each site)
* Any Axis I Psychiatric Disorder as assessed by the MINI that is significantly impairing and/or would contraindicate participation in the study
* Psychiatric medication changes in the past 3 months including new prescriptions, changes in dosages or discontinuation of medications
* Positive toxicology screen for any of the following drugs: cocaine, opiates, methadone, benzodiazepines, barbiturates, amphetamines, methamphetamines, and PCP (Marijuana will be tested for but will not be an exclusionary criterion, participants with valid prescriptions for opiates, benzodiazepines, barbiturates, amphetamines or methadone will not be excluded, participants failing the toxicology screen will be allowed to re-screen once. These participants will need to be re-consented before being rescreened to ensure they have received adequate informed consent.)
* Breath alcohol level > 0.01 (Participants failing the breath alcohol screen will be allowed to re-screen once. These participants will need to be re-consented before being rescreened to ensure they have received adequate informed consent.)
* Current diagnosis of DSM alcohol or drug use disorder (except for nicotine)
* Pregnant, trying to become pregnant or breastfeeding
* Smoking 'roll your own cigarettes' exclusively
* Currently taking anticonvulsant medications including: Phenytoin [Brand Name: Dilantin], Carbamazepine [Brand Name: Tegretol, Carbatrol, Equetro, Epitol], Oxcarbazepine [Brand Name: Trileptal], Primidone [Brand Name: Mysoline], Phenobarbital
* CO reading >80 ppm
* Systolic BP between 90 and 160 (If below 90 then asymptomatic. Participants failing for blood pressure will be allowed to re-screen once.)
* Diastolic BP between 50 and 100 (If below 50 then asymptomatic. Participants failing for blood pressure will be allowed to re-screen once.)
* Heart rate between 45 and 115 bpm (If below 45 then asymptomatic. Participants failing for heart rate will be allowed to re-screen once.)
* Indicating any suicidal ideation in the past month or suicide attempts in the past 10 years.
* Inability to independently read and comprehend the consent form and other written study materials and measures.
* Having participated in a research study during the past three months in which the participant: Smoked a cigarette that was not his/her usual brand cigarette for more than one day, used any tobacco products beyond normal use for more than one day, used any nicotine replacement products or smoking cessation medications for more than one day
* Any previous experience using SPECTRUM cigarettes

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2016-03-30 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-09-12 (Actual)

PRIMARY OUTCOMES:
Number of cigarettes smoked per day | Six weeks
  Self-reported number of cigarettes smoked per day
Composite measure of influence of reduced nicotine content on ADHD symptoms measured by ADHD Rating Scale and Clinical Global Impressions Scale along with related measures of cognition measured by the N-Back Task and the Continuous Performance Test | Six weeks
  Composite of ADHD symptom questionnaires, inhibitory control, working memory
Composite measure of outcomes associated with acceptability; withdrawal measured by the MNWS and compliance measured by Time-Line Follow-Back questionnaire and daily self-report cigarette use | Six weeks
  Composite of study dropout, compliance, changes in physical health

SECONDARY OUTCOMES:
Measures of discomfort/dysfunction; withdrawal and depression | Six weeks
  Withdrawal scale and depression measures
Measures of other health-related behaviors; dependence measures | Six weeks
  Drug and alcohol use questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kollins, Ph.D., Principal Investigator — Duke ADHD Program
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania